CLINICAL TRIAL: NCT06020027
Title: Water is K'é: Multi-level Intervention to Promote Healthy Beverage Choices Among Navajo Families
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California Nutrition Policy Institute (Unknown); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Sonya Sunhi Shin, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023P002075
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Water; Child Nutrition; Family Dynamics; Healthy Nutrition; Healthy Lifestyle; Health-Related Behavior; Obesity Prevention
Keywords: community; Navajo; indigenous; early child health; cultural intervention; family-based intervention; beverage consumption; sugar-sweetened beverages
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Water is K'é is an early child education (ECE) intervention designed to promote family-centered choice using a strength-based approach. Water is K'é promotes multilevel change through strengthened cultural connections, enhanced health literacy, and increased access to drinking water, with the goal of promoting family cohesion and improving health outcomes among family members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Water is K'é is a family-based intervention aimed at improving health and wellness of family members and of the family as a whole. The multi-level intervention targets change at environmental, community and family levels through three core activities: a lesson plan, social media campaign and water access plan. ECE staff will receive a brief training on the curriculum and its relation to the Navajo Wellness Model before delivering the lessons and posting messages. Four interactive lesson plans will be delivered by ECE staff. Caregiver and family sessions will be delivered at the Head Start / FACE facility or in the home, depending on staff preference.
  Interventions: Behavioral: Water is K'é
- Control Arm (No Intervention): Participants attending an ECE site randomly assigned to "waitlist" will receive usual programs and services at the site.

INTERVENTIONS:
Behavioral: Water is K'é — Four-month multi-level, family-based intervention that is grounded in Navajo culture and promotes individual knowledge, motivation and skills; social norms; and environmental changes (access to drinking water). At minimum, the enrolled child and primary caregiver will attend monthly sessions, with an open invitation to other family members. Families will also receive social media posts and develop a family access plan by selecting strategies (if needed) to boost their confidence in their water sources at home. ECE sites will also develop a tailored access plan, selecting strategies to increase confidence in water offered at the ECE site, and implement their access plan with study team support.
  Other Names: Water is K'e
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to understand if a cultural intervention for Navajo families will improve healthy beverage habits, health outcomes, and family cohesion. The main questions it aims to answer are:

* Does Water is K'é results in healthier beverage habits among children aged 2 to 5, compared with children in a control group?
* Does the intervention improve the health of other family members?
* How does the intervention affect family well-being?

Participants will take part in a four-month program at the early child education site (such as a Head Start or the Bureau of Indian Affair's Family and Child Education or FACE Program) where the child is enrolled. They will take part in lesson plans, a social media campaign, and a family water access plan. Researchers will compare the participating families with families at wait-list early child educations sites. We will collect information through surveys, health measurements, and qualitative interviews and compare results to learn if Water is K'e improves health behaviors, health outcomes, and family cohesion.

DETAILED DESCRIPTION:
Water is K'é is a culturally-grounded, family-based intervention designed to promote healthy beverage consumption among Navajo families. Delivered by early child education (ECE) staff, Water is K'é includes three strategies: promoting Diné (Navajo) culture through intergenerational sharing, increasing health literacy about water and sugar-sweetened beverages (SSBs), and increasing drinking water access in both home and ECE settings. Activities consist of a lesson plan for children and caregivers, a tailored access plan to promote confidence in water quality at home and ECE sites; and a social media campaign. Water is K'é is guided by the conceptual framework of the Navajo Wellness Model, addressing four aspects: spiritual; sustenance; family and kinship (K'é); and the environment. The intervention's goal is to promote healthy behaviors and intergenerational sharing of cultural teachings about water, resulting in better health among family members and greater family cohesion overall.

This prospective cluster-randomized trial evaluates the impact of Water is K'é on healthy beverage consumption, health outcomes, and family cohesion. A total of 25 ECE sites will be enrolled in the study, serving in the waitlist group for one year, and then the intervention group the following year based on random assignment. Stepwise roll-out will ensure adequate bandwidth to support intervention sites, while also gathering control data from waitlist sites. Primary caregivers will consent for themselves and the child who is enrolled in the ECE program; other family members will be invited to enroll in the study as well. Each site will enroll approximately 11 families per year, resulting in a total enrollment of 440 families (220 in the intervention group, 220 in the control group) and follow them for 12 months to evaluate the impact on behaviors (beverage consumption patterns) and health outcomes (body mass index, A1c among adults living with diabetes or pre-diabetes) of children and adults. In addition, convergent parallel mixed methods will be used to explore whether Water is K'é results in greater family cohesion through intergenerational cultural continuity. Specific aims are:

1. Evaluate the impact of Water is K'é on children aged 2 to 5. Hypothesis: participating children will have healthier beverage habits and body mass indices compared with children in the control group.
2. Evaluate intervention impact on the health of other family members. Hypothesis: participating individuals will have healthier beverage habits and body mass indices compared with the control group.
3. Evaluate the intervention's impact on family well-being. Hypothesis: participating families will have stronger family cohesion through strengthening of intergenerational cultural continuity compared with families in the control group.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following: child enrolled in participating early child education (ECE) program between 2 and 5 years of age; primary caregiver of that child (i.e. identifies as the person who assumes primary caregiver responsibilities of and resides in the same household as the child; or family member aged six or older identified by primary caregiver as an individual in the immediate family who either resides in the same household or visits frequently and day to day interactions with child);
* Plans to reside in the same household for the next 12 months
* If enrolled in ECE program, plans to participate in ECE program for the entire school year

Exclusion Criteria:

* Plans to leave their residence in the next 12 months
* If enrolled in ECE program, does not plan to participate in ECE program for the entire school year

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Average daily intake of water (fluid ounces) among ECE children | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences based on Beverage Intake Questionnaire Preschool (BEVQ-PS) measurements in frequency and amount across beverage categories, validated in children under 6
Average daily intake of SSB (fluid ounces) among ECE children | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences per BEVQ-PS measurements frequency and amount by beverage type, validated in children under 6
Average daily energy intake from SSB (in calories) among ECE children | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences per BEVQ-PS; measures frequency and amount by beverage type, validated in children under 6
Average daily intake of water (fluid ounces) among family members | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences per Beverage Intake Questionnaire (BEVQ-15); measures frequency and amount across beverage categories, validated for children 6 and older
Average daily intake of SSB (fluid ounces) among family members | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences per BEVQ-PS; measures frequency and amount by beverage type
Average daily energy intake from SSB (in calories) among family members | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences per BEVQ-PS; measures frequency and amount by beverage type, validated in children under 6
Family cohesion score | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Study arm differences based on 10-question instrument adapted from Family Adaptability and Cohesion Scale, Short Form (FACES-SF) subscale to measure family cohesion; completed by all family members over 12. For each family, scores from all family members will be averaged to derive a single score per family.

SECONDARY OUTCOMES:
Age-adjusted body mass index z-score among ECE children | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Height and weight collected using the National Health and Nutrition Examination Survey (NHANES) protocol
Study arm differences in average World Health Organization-5 (WHO-5) score among family members | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  WHO-5: 5-item questionnaire to measure well-being; range 0 to 2t with higher score reflecting greater wellbeing
Perceived access to drinking water | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Question (Likert score 1-5) on perceived access to reliable drinking water; range 0-5 with higher score reflecting greater access.
Perceived confidence in drinking water | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Question (Likert score 1-5) on confidence in drinking water' range 0-5 with higher score reflecting greater confidence.
Knowledge of traditional teachings related to water | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Question (Likert score 1-5) on knowledge of Navajo culture related to water; range 0-5 with higher score reflecting greater knowledge.
Influence of traditional teaching on beverage choices | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Question (Likert score 1-5) on influence of Navajo culture on what drinks offered to child; range 0-5 with higher score reflecting greater influence.

OTHER OUTCOMES:
Exploratory: Study arm differences in change in glycosylated hemoglobin A1c among individuals living with diabetes or pre-diabetes | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Average value of two A1c measures taken at each time point
Exploratory: Study arm differences in average age-adjusted body mass index z-score among family members | Post intervention (at 4 months) and 8 months after intervention (at 12 months from baseline)
  Height and weight collected using NHANES protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Navajo Nation Head Start, Window Rock, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Per stipulations of the Navajo Research Code, all data belongs to Navajo Nation; researchers would need to direct any request for study data, including IPD, to the Navajo Nation Human Research Review Board